CLINICAL TRIAL: NCT04003844
Title: Multicenter, Single-arm, Phase IV Study to Evaluate the Efficacy, Safety of Combined Therapy of Aspirin and IVIG-SN 10% in Pediatric Patients With Kawasaki Disease
Brief Title: Study of Combined Therapy IVIG-SN 10% and Acetylsalicylic Acid in Kawasaki Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC5107E
Record Dates: First submitted 2019-05-16; First posted 2019-07-01 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Immunoglobulin G; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Investigational product (IP)
  Interventions: Drug: Immunoglobulin G; Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Immunoglobulin G — single dose of IGIV 10% (2 g/kg) administered intravenously for at least 12 hours
Drug: Acetylsalicylic acid — Coadministration

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of high-dose human Immunoglobulin G Intravenous (IGIV) 10% in subjects with Kawasaki diseases (KD).

DETAILED DESCRIPTION:
This is a multicenter, single-arm, and open-label clinical trial to evaluate the coronary artery lesions (CALs) at 2 and 7 weeks after single dose of IGIV 10% (2 g/kg) administration for at least 12 hours to evaluate the efficacy and safety of IGIV 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and children aged 3 months to 7 years inclusive, at the time of signing the informed consent, however, patients with complete KD are eligible up to 12 years (applies to 2A)
2. Subjects with fever 4-10 days meeting one of following criteria (A, B or C)

   A. Subjects with at least 4 of the following principal clinical findings:

   i) Bilateral bulbar conjunctival injection without exudate

   ii) Erythema and cracking of lips, strawberry tongue, and/or erythema of oral and pharyngeal mucosa

   iii) Erythema and edema of the hands and feet in acute phase and/or periungual desquamation in subacute phase

   iv) Cervical lymphadenopathy (≥1.5 cm diameter), usually unilateral

   v) Rash: maculopapular, diffuse erythroderma, or erythema multiforme-like

   B. Subjects with at least 3 of the principal clinical findings and coronary artery abnormalities detected by 2-dimensional echocardiography: Z score of left anterior descending coronary artery or right coronary artery ≥2.5

   C. Subjects without coronary artery abnormalities, but with fever ≥5 days, 2 or 3 of the principal clinical findings , CRP of ≥3.0 mg/dL and meeting 3 or more of the following laboratory findings:

   i) Albumin <3.0 g/dL

   ii) Anemia for age

   iii) Elevated alanine aminotransferase level

   iv) Platelet count of >450,000/mm3 after the 7th day of fever

   v) White blood cell count of >15,000/mm3

   vi) Urine >10 white blood cells/high-power field
3. Subjects whose subject's parents or legally authorized representative gave voluntary written consent to participate in the clinical trial

Exclusion Criteria:

1. Subjects with a history of KD
2. Subjects with following laboratory findings:

   A. Platelet count <100,000/mm3

   B. WBC count <3,000 cells/mm3

   C. hemoglobin, hematocrit or red blood cell count more than 30% above the upper limit or 30% below the lower limit of the normal range
3. Subjects who are currently receiving or who have received any investigational drug or device within 30 days prior to administration of the IP
4. Subjects who have received TNF alpha antagonist or systemic corticosteroids within 48 hours prior to administration of the IP
5. Subjects who are considered by the investigator to be an unsuitable candidate for the study due to a severe chronic disease (e.g. cardiovascular disease except controllable hypertension, respiratory disease with respiratory failure, metabolic disease, renal failure, hemoglobinopathy, etc.)
6. Subjects who have received immunosuppressive or immunomodulatory drugs within 3 months prior to administration of the IP
7. Subjects with immunodeficiency including known positive serology for human immunodeficiency virus (HIV)
8. Subjects with a history of hypersensitivity or shock to IVIG formulations
9. Subjects with underlying liver disease or liver dysfunction with known etiology
10. Subjects with renal impairment whose creatinine level is more than twice the upper limit of the normal range
11. Subjects with a history of malignant tumor
12. Subjects with a history of IgA deficiency
13. Subjects who are considered by the investigator to be an unsuitable candidate for the study for any reason

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
incidence of CALs | 7 weeks
  incidence of CALs at 7 weeks after treatment

SECONDARY OUTCOMES:
incidence of CALs | 2 weeks
  incidence of CALs at 2 weeks after treatment
total duration of fever | baseline
  total duration of fever after treatment
laboratory measurements : markers of inflammation and cardiovascular disease | 7 weeks
  measurement of erythrocyte sedimentation rate (ESR)
laboratory measurements : markers of inflammation and cardiovascular disease | 7 weeks
  measurement of C-reactive protein (CRP)
laboratory measurements : markers of inflammation and cardiovascular disease | 7 weeks
  measurement of N-terminal pro B-type natriuretic peptide (NTproBNP) or B-type natriuretic peptide (BNP)
laboratory measurements : markers of inflammation and cardiovascular disease | 7 weeks
  measurement of creatine kinase-myocardial band (CK-MB)
laboratory measurements : markers of inflammation and cardiovascular disease | 7 weeks
  measurement of procalcitonin
laboratory measurements : markers of inflammation and cardiovascular disease | 7 weeks
  measurement of soluble suppression of tumorigenicity 2 (sST2)
laboratory measurements : markers of inflammation and cardiovascular disease | 7 weeks
  measurement of Troponin I
IGIV resistance | baseline
  frequency of IGIV resistance
adverse events, adverse drug reactions and serious adverse events | 7 weeks
  number of adverse events, adverse drug reactions and serious adverse events
laboratory measurements : hematological parameters | 7 weeks
  measurement of white blood cell (WBC)
laboratory measurements : hematological parameters | 7 weeks
  measurement of red blood cell (RBC)
laboratory measurements : hematological parameters | 7 weeks
  measurement of hemoglobin
laboratory measurements : hematological parameters | 7 weeks
  measurement of hematocrit
laboratory measurements : hematological parameters | 7 weeks
  measurement of platelet count
laboratory measurements : clinical chemistry parameters | 7 weeks
  measurement of alanine transaminase (ALT)
laboratory measurements : clinical chemistry parameters | 7 weeks
  measurement of albumin
laboratory measurements : urinalysis | 7 weeks
  measurement of WBC (urine microscopy)
vital signs: blood pressure | 7 weeks
  measurement of systolic and diastolic blood pressure
vital signs: body temperature | 7 weeks
  measurement of body temperature
physical examination | 7 weeks
  visual inspection of general appearance, head, eyes, nose-mouth-throat, lymph nodes, skin, extremities for abnormal findings

CONTACTS AND LOCATIONS:
Overall Officials: Mi Young Han, MD, Ph.D., Principal Investigator — Kyunghee University Medical Center
Locations (7):
- South Korea (7):
  - Hallym University Sacred Heart Hospital, Anyang
  - Asan Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju